CLINICAL TRIAL: NCT03092479
Title: A Randomized Trial of a Pilot Behavioral Support Intervention After Bariatric Surgery
Brief Title: Pilot Behavioral Support Intervention After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-0469
Record Dates: First submitted 2017-03-15; First posted 2017-03-28 (Actual); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention (Experimental): 4-month bi-weekly comprehensive postoperative behavioral support program addressing psychosocial changes after surgery, strategies for postoperative diet and adherence and preventing weight regain.
  Interventions: Behavioral: Behavioral Intervention
- Usual Care (No Intervention): Usual postoperative follow-up per the GHS Center for Nutrition and Weight Management guidelines.

INTERVENTIONS:
Behavioral: Behavioral Intervention — Eight bi-weekly small group sessions of approximately 10 participants with session content focused on addressing psychosocial changes after surgery, strategies for postoperative diet and adherence and preventing weight regain.
  Arms: Behavioral Intervention

SUMMARY:
Prospective, randomized pilot trial to evaluate a comprehensive postoperative behavioral support intervention using a 4-month bi-weekly program in 40 bariatric surgery patients (all surgical procedure types) from the Geisinger Health System Center for Nutrition and Weight Management compared to 40 usual care patients.

DETAILED DESCRIPTION:
Bariatric surgery patients may experience significant psychosocial changes after surgery, but little psychological support is available beyond support groups postoperatively. Psychosocial changes after surgery, including mood fluctuations, interpersonal issues and substance use, have the potential to lower quality of life and interfere with adherence to the postoperative diet and lifestyle, diminishing weight loss outcomes.

This prospective randomized pilot trial will evaluate the effect of a postoperative support program targeting quality of life, psychosocial functioning and adherence to behavior change in Geisinger Health System (GHS) bariatric surgery patients.

In this study there will be two arms. The intervention arm will include forty bariatric surgery patients (all procedure types) from the GHS Center for Nutrition and Weight Management (CNWM) who will participate in a four month bi-weekly postoperative behavioral support program to address psychosocial changes after surgery, strategies for postoperative diet and adherence and preventing weight regain. The control arm will include 40 usual care (UC) patients from the same center that completed bariatric surgery within one year.

Both groups will complete two sets of surveys. The first set will be administered at study initiation. The second set will be administered upon completion of the 8 sessions for the intervention group. The control group will also complete surveys during this same timeframe (approximately 4-6 months after baseline survey completion).

Upon study completion, control group members will be afforded an opportunity to participate in the same postoperative behavioral support program offered to the intervention group.

The primary endpoint of this study will be quality of life with secondary endpoints including differences in psychosocial functioning (mood, eating behaviors) and adherence (diet, physical activity, appointments) as well as patient satisfaction, treatment feasibility and attrition.

ELIGIBILITY:
Inclusion Criteria:

* BMI>35 kg/m2 at time of surgery
* Primary bariatric surgery completion < 1 year
* Understanding of informed consent

Exclusion Criteria:

* Pregnancy
* Revision of bariatric surgery
* Significant cognitive impairment that prevents informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Campbell, PhD, Principal Investigator — Geisinger Clinic; Michelle Lent, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Courcoulas AP, Christian NJ, Belle SH, Berk PD, Flum DR, Garcia L, Horlick M, Kalarchian MA, King WC, Mitchell JE, Patterson EJ, Pender JR, Pomp A, Pories WJ, Thirlby RC, Yanovski SZ, Wolfe BM; Longitudinal Assessment of Bariatric Surgery (LABS) Consortium. Weight change and health outcomes at 3 years after bariatric surgery among individuals with severe obesity. JAMA. 2013 Dec 11;310(22):2416-25. doi: 10.1001/jama.2013.280928. PMID 24189773
- [Background] Mechanick JI, Youdim A, Jones DB, Garvey WT, Hurley DL, McMahon MM, Heinberg LJ, Kushner R, Adams TD, Shikora S, Dixon JB, Brethauer S; American Association of Clinical Endocrinologists; Obesity Society; American Society for Metabolic & Bariatric Surgery. Clinical practice guidelines for the perioperative nutritional, metabolic, and nonsurgical support of the bariatric surgery patient--2013 update: cosponsored by American Association of Clinical Endocrinologists, The Obesity Society, and American Society for Metabolic & Bariatric Surgery. Obesity (Silver Spring). 2013 Mar;21 Suppl 1(0 1):S1-27. doi: 10.1002/oby.20461. PMID 23529939
- [Background] Livhits M, Mercado C, Yermilov I, Parikh JA, Dutson E, Mehran A, Ko CY, Gibbons MM. Preoperative predictors of weight loss following bariatric surgery: systematic review. Obes Surg. 2012 Jan;22(1):70-89. doi: 10.1007/s11695-011-0472-4. PMID 21833817
- [Background] Herpertz S, Kielmann R, Wolf AM, Hebebrand J, Senf W. Do psychosocial variables predict weight loss or mental health after obesity surgery? A systematic review. Obes Res. 2004 Oct;12(10):1554-69. doi: 10.1038/oby.2004.195. PMID 15536219
- [Background] Bauchowitz AU, Gonder-Frederick LA, Olbrisch ME, Azarbad L, Ryee MY, Woodson M, Miller A, Schirmer B. Psychosocial evaluation of bariatric surgery candidates: a survey of present practices. Psychosom Med. 2005 Sep-Oct;67(5):825-32. doi: 10.1097/01.psy.0000174173.32271.01. PMID 16204445
- [Background] King WC, Chen JY, Mitchell JE, Kalarchian MA, Steffen KJ, Engel SG, Courcoulas AP, Pories WJ, Yanovski SZ. Prevalence of alcohol use disorders before and after bariatric surgery. JAMA. 2012 Jun 20;307(23):2516-25. doi: 10.1001/jama.2012.6147. PMID 22710289
- [Background] Sarwer DB, Wadden TA, Fabricatore AN. Psychosocial and behavioral aspects of bariatric surgery. Obes Res. 2005 Apr;13(4):639-48. doi: 10.1038/oby.2005.71. PMID 15897471
- [Background] Tindle HA, Omalu B, Courcoulas A, Marcus M, Hammers J, Kuller LH. Risk of suicide after long-term follow-up from bariatric surgery. Am J Med. 2010 Nov;123(11):1036-42. doi: 10.1016/j.amjmed.2010.06.016. Epub 2010 Sep 16. PMID 20843498
- [Background] Bradley LE, Sarwer DB, Forman EM, Kerrigan SG, Butryn ML, Herbert JD. A Survey of Bariatric Surgery Patients' Interest in Postoperative Interventions. Obes Surg. 2016 Feb;26(2):332-8. doi: 10.1007/s11695-015-1765-9. PMID 26084251
- [Background] Puzziferri N, Roshek TB 3rd, Mayo HG, Gallagher R, Belle SH, Livingston EH. Long-term follow-up after bariatric surgery: a systematic review. JAMA. 2014 Sep 3;312(9):934-42. doi: 10.1001/jama.2014.10706. PMID 25182102
- [Background] Adams TD, Davidson LE, Litwin SE, Kolotkin RL, LaMonte MJ, Pendleton RC, Strong MB, Vinik R, Wanner NA, Hopkins PN, Gress RE, Walker JM, Cloward TV, Nuttall RT, Hammoud A, Greenwood JL, Crosby RD, McKinlay R, Simper SC, Smith SC, Hunt SC. Health benefits of gastric bypass surgery after 6 years. JAMA. 2012 Sep 19;308(11):1122-31. doi: 10.1001/2012.jama.11164. PMID 22990271
- [Background] Pekkarinen T, Koskela K, Huikuri K, Mustajoki P. Long-term Results of Gastroplasty for Morbid Obesity: Binge-Eating as a Predictor of Poor Outcome. Obes Surg. 1994 Aug;4(3):248-255. doi: 10.1381/096089294765558467. PMID 10742782
- [Background] DiMatteo MR, Lepper HS, Croghan TW. Depression is a risk factor for noncompliance with medical treatment: meta-analysis of the effects of anxiety and depression on patient adherence. Arch Intern Med. 2000 Jul 24;160(14):2101-7. doi: 10.1001/archinte.160.14.2101. PMID 10904452
- [Background] Piette JD, Heisler M, Ganoczy D, McCarthy JF, Valenstein M. Differential medication adherence among patients with schizophrenia and comorbid diabetes and hypertension. Psychiatr Serv. 2007 Feb;58(2):207-12. doi: 10.1176/ps.2007.58.2.207. PMID 17287377
- [Background] Kinzl JF, Schrattenecker M, Traweger C, Mattesich M, Fiala M, Biebl W. Psychosocial predictors of weight loss after bariatric surgery. Obes Surg. 2006 Dec;16(12):1609-14. doi: 10.1381/096089206779319301. PMID 17217637
- [Background] Clark MM, Balsiger BM, Sletten CD, Dahlman KL, Ames G, Williams DE, Abu-Lebdeh HS, Sarr MG. Psychosocial factors and 2-year outcome following bariatric surgery for weight loss. Obes Surg. 2003 Oct;13(5):739-45. doi: 10.1381/096089203322509318. PMID 14627469
- [Background] Thonney B, Pataky Z, Badel S, Bobbioni-Harsch E, Golay A. The relationship between weight loss and psychosocial functioning among bariatric surgery patients. Am J Surg. 2010 Feb;199(2):183-8. doi: 10.1016/j.amjsurg.2008.12.028. Epub 2009 Apr 10. PMID 19362287
- [Background] Sarwer DB, Cohn NI, Gibbons LM, Magee L, Crerand CE, Raper SE, Rosato EF, Williams NN, Wadden TA. Psychiatric diagnoses and psychiatric treatment among bariatric surgery candidates. Obes Surg. 2004 Oct;14(9):1148-56. doi: 10.1381/0960892042386922. PMID 15527626
- [Background] Allison KC, Wadden TA, Sarwer DB, Fabricatore AN, Crerand CE, Gibbons LM, Stack RM, Stunkard AJ, Williams NN. Night eating syndrome and binge eating disorder among persons seeking bariatric surgery: prevalence and related features. Obesity (Silver Spring). 2006 Mar;14 Suppl 2:77S-82S. doi: 10.1038/oby.2006.286. PMID 16648598
- [Background] Rudolph A, Hilbert A. Post-operative behavioural management in bariatric surgery: a systematic review and meta-analysis of randomized controlled trials. Obes Rev. 2013 Apr;14(4):292-302. doi: 10.1111/obr.12013. Epub 2013 Jan 7. PMID 23294936
- [Background] Kolotkin RL, Meter K, Williams GR. Quality of life and obesity. Obes Rev. 2001 Nov;2(4):219-29. doi: 10.1046/j.1467-789x.2001.00040.x. PMID 12119993
- [Background] Libeton M, Dixon JB, Laurie C, O'Brien PE. Patient motivation for bariatric surgery: characteristics and impact on outcomes. Obes Surg. 2004 Mar;14(3):392-8. doi: 10.1381/096089204322917936. PMID 15072662
- [Background] Goldman RL, Borckardt JJ, Frohman HA, O'Neil PM, Madan A, Campbell LK, Budak A, George MS. Prefrontal cortex transcranial direct current stimulation (tDCS) temporarily reduces food cravings and increases the self-reported ability to resist food in adults with frequent food craving. Appetite. 2011 Jun;56(3):741-6. doi: 10.1016/j.appet.2011.02.013. Epub 2011 Feb 23. PMID 21352881
- [Background] Lent MR, Hayes SM, Wood GC, Napolitano MA, Argyropoulos G, Gerhard GS, Foster GD, Still CD. Smoking and alcohol use in gastric bypass patients. Eat Behav. 2013 Dec;14(4):460-3. doi: 10.1016/j.eatbeh.2013.08.008. Epub 2013 Aug 17. PMID 24183136
- [Background] Lent MR, Napolitano MA, Wood GC, Argyropoulos G, Gerhard GS, Hayes S, Foster GD, Collins CA, Still CD. Internalized weight bias in weight-loss surgery patients: psychosocial correlates and weight loss outcomes. Obes Surg. 2014 Dec;24(12):2195-9. doi: 10.1007/s11695-014-1455-z. PMID 25337868
- [Background] Hayes S, Napolitano MA, Lent MR, Wood GC, Gerhard GS, Irving BA, Argyropoulos G, Foster GD, Still CD. The effect of insurance status on pre- and post-operative bariatric surgery outcomes. Obes Surg. 2015 Jan;25(1):191-4. doi: 10.1007/s11695-014-1478-5. PMID 25373925
- [Background] Hirsch AG, Wood GC, Bailey-Davis L, Lent MR, Gerhard GS, Still CD. Collateral weight loss in children living with adult bariatric surgery patients: a case control study. Obesity (Silver Spring). 2014 Oct;22(10):2224-9. doi: 10.1002/oby.20827. Epub 2014 Jul 2. PMID 24989939
- [Background] Lent MR, Swencionis C. Addictive personality and maladaptive eating behaviors in adults seeking bariatric surgery. Eat Behav. 2012 Jan;13(1):67-70. doi: 10.1016/j.eatbeh.2011.10.006. Epub 2011 Oct 20. PMID 22177401
- [Background] Kofman MD, Lent MR, Swencionis C. Maladaptive eating patterns, quality of life, and weight outcomes following gastric bypass: results of an Internet survey. Obesity (Silver Spring). 2010 Oct;18(10):1938-43. doi: 10.1038/oby.2010.27. Epub 2010 Feb 18. PMID 20168309
- [Background] Still CD, Benotti P, Wood GC, Gerhard GS, Petrick A, Reed M, Strodel W. Outcomes of preoperative weight loss in high-risk patients undergoing gastric bypass surgery. Arch Surg. 2007 Oct;142(10):994-8; discussion 999. doi: 10.1001/archsurg.142.10.994. PMID 17938314
- [Background] Still CD, Wood GC, Chu X, Manney C, Strodel W, Petrick A, Gabrielsen J, Mirshahi T, Argyropoulos G, Seiler J, Yung M, Benotti P, Gerhard GS. Clinical factors associated with weight loss outcomes after Roux-en-Y gastric bypass surgery. Obesity (Silver Spring). 2014 Mar;22(3):888-94. doi: 10.1002/oby.20529. Epub 2014 Feb 6. PMID 23804287
- [Background] Wood GC, Chu X, Manney C, Strodel W, Petrick A, Gabrielsen J, Seiler J, Carey D, Argyropoulos G, Benotti P, Still CD, Gerhard GS. An electronic health record-enabled obesity database. BMC Med Inform Decis Mak. 2012 May 28;12:45. doi: 10.1186/1472-6947-12-45. PMID 22640398
- [Background] Berkowitz RI. Treating Adolescent Obesity. Adolesc Med. 1997 Feb;8(1):181-195. PMID 10360016
- [Background] McHorney CA, Ware JE Jr, Lu JF, Sherbourne CD. The MOS 36-item Short-Form Health Survey (SF-36): III. Tests of data quality, scaling assumptions, and reliability across diverse patient groups. Med Care. 1994 Jan;32(1):40-66. doi: 10.1097/00005650-199401000-00004. PMID 8277801
- [Background] Jenkinson C, Wright L, Coulter A. Criterion validity and reliability of the SF-36 in a population sample. Qual Life Res. 1994 Feb;3(1):7-12. doi: 10.1007/BF00647843. PMID 8142947
- [Background] Wee CC, Davis RB, Hamel MB. Comparing the SF-12 and SF-36 health status questionnaires in patients with and without obesity. Health Qual Life Outcomes. 2008 Jan 30;6:11. doi: 10.1186/1477-7525-6-11. PMID 18234099
- [Background] Doll HA, Petersen SE, Stewart-Brown SL. Obesity and physical and emotional well-being: associations between body mass index, chronic illness, and the physical and mental components of the SF-36 questionnaire. Obes Res. 2000 Mar;8(2):160-70. doi: 10.1038/oby.2000.17. PMID 10757202
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Pinaquy S, Chabrol H, Simon C, Louvet JP, Barbe P. Emotional eating, alexithymia, and binge-eating disorder in obese women. Obes Res. 2003 Feb;11(2):195-201. doi: 10.1038/oby.2003.31. PMID 12582214
- [Background] Paffenbarger RS Jr, Wing AL, Hyde RT. Physical activity as an index of heart attack risk in college alumni. 1978. Am J Epidemiol. 1995 Nov 1;142(9):889-903; discussion 887-8. doi: 10.1093/oxfordjournals.aje.a117736. No abstract available. PMID 7572969
- [Background] Bond DS, Jakicic JM, Unick JL, Vithiananthan S, Pohl D, Roye GD, Ryder BA, Sax HC, Wing RR. Pre- to postoperative physical activity changes in bariatric surgery patients: self report vs. objective measures. Obesity (Silver Spring). 2010 Dec;18(12):2395-7. doi: 10.1038/oby.2010.88. Epub 2010 Apr 8. PMID 20379143
- [Background] Latner JD, Mond JM, Kelly MC, Haynes SN, Hay PJ. The Loss of Control Over Eating Scale: development and psychometric evaluation. Int J Eat Disord. 2014 Sep;47(6):647-59. doi: 10.1002/eat.22296. Epub 2014 May 26. PMID 24862351
- [Background] Arnow B, Kenardy J, Agras WS. The Emotional Eating Scale: the development of a measure to assess coping with negative affect by eating. Int J Eat Disord. 1995 Jul;18(1):79-90. doi: 10.1002/1098-108x(199507)18:13.0.co;2-v. PMID 7670446
- [Background] Weissman MM, Bothwell S. Assessment of social adjustment by patient self-report. Arch Gen Psychiatry. 1976 Sep;33(9):1111-5. doi: 10.1001/archpsyc.1976.01770090101010. PMID 962494
- [Background] Weissman MM, Prusoff BA, Thompson WD, Harding PS, Myers JK. Social adjustment by self-report in a community sample and in psychiatric outpatients. J Nerv Ment Dis. 1978 May;166(5):317-26. doi: 10.1097/00005053-197805000-00002. PMID 650195
- [Background] Sarwer DB, Wadden TA, Moore RH, Baker AW, Gibbons LM, Raper SE, Williams NN. Preoperative eating behavior, postoperative dietary adherence, and weight loss after gastric bypass surgery. Surg Obes Relat Dis. 2008 Sep-Oct;4(5):640-6. doi: 10.1016/j.soard.2008.04.013. Epub 2008 Jun 30. PMID 18586571
- [Background] Sarwer DB, Moore RH, Spitzer JC, Wadden TA, Raper SE, Williams NN. A pilot study investigating the efficacy of postoperative dietary counseling to improve outcomes after bariatric surgery. Surg Obes Relat Dis. 2012 Sep-Oct;8(5):561-8. doi: 10.1016/j.soard.2012.02.010. Epub 2012 Mar 21. PMID 22551576
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] de Zwaan M, Lancaster KL, Mitchell JE, Howell LM, Monson N, Roerig JL, Crosby RD. Health-related quality of life in morbidly obese patients: effect of gastric bypass surgery. Obes Surg. 2002 Dec;12(6):773-80. doi: 10.1381/096089202320995547. PMID 12568181
- [Background] Hollis S. A graphical sensitivity analysis for clinical trials with non-ignorable missing binary outcome. Stat Med. 2002 Dec 30;21(24):3823-34. doi: 10.1002/sim.1276. PMID 12483769
- [Background] Spielberger CD. State-trait anxiety inventory: a comprehensive bibliography. 2nd ed. Palo Alto, CA: Consulting Psychologists Press; 1989.
- [Background] Clark MM, Abrams DB, Niaura RS, Eaton CA, Rossi JS. Self-efficacy in weight management. J Consult Clin Psychol. 1991 Oct;59(5):739-44. doi: 10.1037//0022-006x.59.5.739. PMID 1955608
- [Background] Edwards DW, Yarvis RM, Mueller DP, Zingale HC, Wagman WJ. Test-Taking and the Stability of Adjustment Scales Can We Assess Patient Deterioration? Evaluation Review 1978;2:275-91.
- [Background] Rubin DB. Multiple Imputation for Nonresponse in Surveys. New York: Wiley and Sons; 1987.
- [Derived] Lent MR, Campbell LK, Kelly MC, Lawson JL, Murakami JM, Gorrell S, Wood GC, Yohn MM, Ranck S, Petrick AT, Cunningham K, LaMotte ME, Still CD. The feasibility of a behavioral group intervention after weight-loss surgery: A randomized pilot trial. PLoS One. 2019 Oct 21;14(10):e0223885. doi: 10.1371/journal.pone.0223885. eCollection 2019. PMID 31634365

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Behavioral Intervention | Usual Care
Started | 24 | 26
Completed | 17 | 24
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Intervention | Usual Care | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (9.1) | 46.2 (12.0) | 46.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 23 | 25 | 48
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 47.1 (6.7) | 50.4 (6.2) | 48.8 (6.6)
Surgery Type [Number; unit: participants]
  RYGB | 17 | 16 | 33
  SG | 7 | 7 | 14
  PD/DS | 0 | 3 | 3
Initial Psychosocial Clearance Light [Number; unit: participants] — Green = cleared for surgery Yellow = delayed clearance and behavioral goals
  participants
    Green | 13 | 15 | 28
    Yellow | 11 | 11 | 22
Months from Surgery to Enrollment [Mean (Standard Deviation); unit: Months] | 7.0 (3.6) | 6.9 (4.1) | 7.0 (3.8)
Baseline Questionnaire Scores - Quality of Life [Mean (Standard Deviation); unit: units on a scale] — Short form-36 (SF-36) has eight quality of life scales that are scored on a range of 0-100 where a higher score indicates a better outcome.
  Loss of control over eating scale-brief (LOCES) is a seven-item measure that is scored on a range of 5-35; higher scores indicate a worse outcome.
  Weight efficacy life-style (WEL, Short Form) is an eight-item measure that is scored on a range of 0-80l higher scores indicate a better outcome.
  units on a scale
    SF-36 Overall | 70.4 (17.9) | 63.3 (18.9) | 66.6 (18.6)
    LOCES | 11.1 (4.1) | 13.0 (5.3) | 12.1 (4.8)
    WELSF | 59.3 (15.8) | 59.0 (17.4) | 59.1 (16.5)
Baseline Questionnaire Scores - Mental Health [Mean (Standard Deviation); unit: units on a scale] — Patient health questionnaire-9 (PHQ-9) is scored on a range of 0-27 where higher scores indicate worse outcomes (scores of five = mild depression, ten = moderate, and fifteen or more = severe); where higher scores indicate a worse outcome. State-trait anxiety inventory (STAI) is a forty-item measure that is scored on a four-point Likert scale of 20-80 per subtest; used for both the State-trait anxiety inventory-state (STAI-S) and State-trait anxiety inventory-trait (STAI-T) where higher scores for both indicate a worse outcome.
  units on a scale
    PHQ-9 | 5.5 (4.5) | 7.5 (5.8) | 6.5 (5.3)
    STAI-S | 45.0 (5.5) | 44.6 (6.1) | 44.8 (5.8)
    STAI-T | 45.7 (6.4) | 45.2 (6.1) | 45.4 (5.4)
Baseline Questionnaire Scores - EES [Mean (Standard Deviation); unit: units on a scale] — Emotional eating scale (EES) is a twenty-five item scale that is scored on two subscale ranges of 0-36 or 0-44; higher scores indicate worse outcomes. This same scale was used across all subsections: EES-Frustration, EES-Anxiety, and EES-Depression. These subscales are reported separately.
  units on a scale
    EES-Frustration | 8.2 (8.1) | 8.5 (8.8) | 8.4 (8.4)
    EES-Anxiety | 8.4 (6.6) | 6.8 (6.8) | 7.6 (6.7)
    EES-Depression | 5.6 (3.9) | 5.5 (4.8) | 5.6 (4.4)
Baseline Questionnaire Scores - Diet and Exercise [Mean (Standard Deviation); unit: units on a scale] — Dietary adherence was measured by a nine-point Likert scale where it was scored on a scale of 1-9; higher scores indicate a better outcome.
  The Paffenbarger Physical Activity Questionnaire (PPAQ) is an eight-item questionnaire that is scored by measuring minutes per week of Moderate to Vigorous Physical Activity (MVPA) by adding block per day and and physical activity of at least moderate level; not measured on a scale.
  units on a scale
    Dietary Adherence | 7.1 (1.3) | 7.4 (1.2) | 7.3 (1.3)
    PPAQ (MVPA min/week) | 120.8 (177) | 82.3 (135) | 100.4 (155)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Mean Health-Related Quality of Life (HRQoL) Scores Related to Physical Function, Energy Level and General Health.
Description: Health-Related Quality of Life emotional scale scores will be assessed by the SF-36-Item Short Form Health Survey between the Behavior Intervention and Control groups. This study seeks a difference of 2/3 standard deviation in scores between groups for statistical significance. Range 0-100. Higher score indicates a better outcome.
Time Frame: Surveys will be completed at baseline and at the completion of the 4 month session time period. Surveys will be provided to both study groups in parallel for consistency.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Intervention | Usual Care
Number analyzed (Participants) | 17 | 24
score on a scale | 11.4 (15.4) | 4.6 (12.1)

2. Secondary Outcome: Difference Between Groups in Depression Scores.
Description: Difference in depression scores between the Behavior Intervention and Control groups will be measured using the total score generated from the Patient Health Questionnaire (PHQ-9). Range is 0-27. Higher score means a worse outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Intervention | Usual Care
Number analyzed (Participants) | 17 | 24
score on a scale | -0.9 (4.6) | -1.1 (4.5)

3. Secondary Outcome: Difference Between Groups in Anxiety Scores.
Description: Difference in anxiety weighted scores between the Behavior Intervention and Control groups will be measured using the scores generated from the State-Trait Anxiety Inventory (STAI) and is scored on a four-point Likert scale. Range is 20-80 per subtest. Higher scores indicate a worse outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Intervention | Usual Care
Number analyzed (Participants) | 17 | 24
units on a scale
  STAI-S | 0.9 (4.9) | 0.3 (6.0)
  STAI-T | -1.5 (4.1) | -0.4 (4.7)

4. Secondary Outcome: Difference Between Groups in Measured Self-efficacy.
Description: Difference in self-efficacy parameters between the Behavior Intervention and Control groups will be measured by comparing responses generated from the Weight Efficacy Life-Style short-form scale (WEL-SF). Range is 0-80. Higher score indicates a better outcome
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Intervention | Usual Care
Number analyzed (Participants) | 17 | 24
score on a scale | 2.0 (14.1) | -1.6 (10.9)

5. Secondary Outcome: Difference in Physical Activity Levels Between Groups.
Description: Differences in physical activity levels between the Behavior Intervention and Control groups will be measured by comparing hours per day spent in vigorous, moderate, light or sitting activity as recorded on the Paffenbarger Physical Activity Questionnaire (PPAQ). Calculated by minutes per week of Moderate to Vigorous Activity (MVPA).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes (min)
Arm/Group | Behavioral Intervention | Usual Care
Number analyzed (Participants) | 17 | 24
minutes (min) | 71 (160) | -14 (145)

6. Secondary Outcome: Difference in Emotional Eating Scale Results Between Groups.
Description: The Emotional Eating scale (EES) measures a subject's desire to eat in response to an emotional stimulus. This scale will be used to assess differences in emotional eating habits between the Behavior Intervention and Control groups. Subscale scores range 0-36 or 0-44. Higher scores indicates worse outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Intervention | Usual Care
Number analyzed (Participants) | 17 | 24
score on a scale
  EES-Frustration | 1.5 (7.1) | 0.1 (7.3)
  EES-Anxiety | -0.4 (7.0) | 1.9 (6.1)
  EES-Depression | 1.5 (4.8) | 0.0 (3.8)

7. Secondary Outcome: Differences Between Groups in Loss of Eating Control.
Description: The Loss of Control Over Eating Scale-Brief (LOCES) provides a 5 point scoring system to assess subject's loss of eating control. This scale will be used to assess differences in this measure between the Behavior Intervention and Control groups. Range is 5-35. Higher score indicates a worse outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Intervention | Usual Care
Number analyzed (Participants) | 17 | 24
score on a scale | 0.1 (3.9) | -0.7 (3.5)

ADVERSE EVENTS:
Time Frame: 16 weeks during behavioral intervention or between first and final questionnaire completion for the usual care arm.
Arm/Group | Behavioral Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26

LIMITATIONS AND CAVEATS:
Under- powered to detect differences between groups and limited to presenting effect sizes only. Cohort was predominantly White, limiting generalizability of our findings. Most study outcomes were self-reported, which can be subject to bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT03092479/Prot_SAP_000.pdf